CLINICAL TRIAL: NCT06926348
Title: Usability, Acceptability, and Preliminary Effectiveness of a Digital Health Technology for Patient Monitoring of Chronic Insomnia Symptoms and the Promotion of Functional Sleep Behaviors: A Randomized Clinical Trial
Brief Title: Assessment of Usability and Preliminary Effectiveness of a Digital Sleep Aid in an Italian Sample
Acronym: REST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Santer Reply S.p.A. Milan, Italy (Unknown); daVi Digital Medicine s.r.l. Verona, Italy (Unknown); QStep s.r.l. Verona, Italy (Unknown); Fondazione RIDE2Med, Milan, Italy (Unknown)
Responsible Party: Principal Investigator, Elena Antelmi, Associate Professor of Neurology and Clinical Neurologist, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 413CET
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Insomnia Chronic; Insomnia
Keywords: Insomnia; CBT-i; Cognitive Behavioral Therapy for Insomnia; Digital Health Technology; DTx
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Digital Health; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Health Technology (DHT) + Treatment As Usual (TAU) (Experimental): Participants in this arm receive an 8-week intervention involving a mobile app designed for chronic insomnia management. The app includes digital sleep diaries, personalized sleep hygiene education, cognitive strategies, relaxation and mindfulness exercises, and an interactive chatbot for enhanced engagement. This intervention complements standard treatment (TAU), which may include pharmacotherapy and routine clinical care.
  Interventions: Behavioral: Digital Health Technology for Chronic Insomnia
- Treatment As Usual (TAU) (Active Comparator): Participants assigned to this arm continue their usual insomnia management, including pharmacological treatments if prescribed, and receive standardized educational material on sleep hygiene practices via a printed booklet. They also maintain printed sleep diaries for self-monitoring throughout the 8-week study period.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Digital Health Technology for Chronic Insomnia — A mobile application designed to support chronic insomnia management through digital self-monitoring of sleep patterns, personalized sleep hygiene education, cognitive strategies, relaxation and mindfulness exercises, and chatbot interactions. Users receive tailored notifications and educational content to encourage healthy sleep behaviors over an 8-week period. Existing pharmacological treatments prescribed prior to study enrollment continue unchanged
  Arms: Digital Health Technology (DHT) + Treatment As Usual (TAU)
Behavioral: Treatment as Usual (TAU) — Participants receive standard sleep hygiene recommendations via a printed educational booklet. They maintain printed sleep diaries for daily self-monitoring throughout the 8-week intervention. Existing pharmacological treatments prescribed prior to study enrollment continue unchanged.
  Arms: Treatment As Usual (TAU)

SUMMARY:
Chronic insomnia affects approximately 30% of the Italian population, leading to significant impairments in daily functioning and overall health. While Cognitive Behavioral Therapy for Insomnia (CBT-I) is the recommended first-line treatment, access is limited due to a shortage of trained specialists and resources within the Italian healthcare system. This study aims to evaluate the usability, acceptability, and preliminary effectiveness of a mobile application designed to assist individuals with chronic insomnia. The app offers digital sleep diaries, personalized sleep hygiene education, relaxation exercises, and an interactive chatbot to promote healthy sleep behaviors. Fifty adult participants diagnosed with chronic insomnia will be randomly assigned to either the intervention group, which will use the mobile application alongside their usual treatment, or to a control group receiving only standard care. The primary outcomes will assess the app's usability and participants' adherence to sleep hygiene practices. Secondary outcomes will evaluate changes in insomnia severity, mood, and quality of life. Assessments will occur at the start of the study, after the 8-week intervention, and at a 6-month follow-up to explore the intervention's long-term effects.

DETAILED DESCRIPTION:
This randomized controlled pilot trial evaluates a Digital Health Technology (DHT) developed as a Health & Wellness tool aimed at supporting individuals diagnosed with chronic insomnia. Chronic insomnia significantly impacts quality of life and poses a considerable burden on healthcare systems. Despite Cognitive Behavioral Therapy for Insomnia (CBT-I) being the recommended first-line treatment, its limited accessibility in Italy necessitates scalable and innovative solutions. The DHT under investigation is a mobile application developed collaboratively by the University of Verona and private-sector partners, designed specifically for educational purposes and the promotion of healthy sleep behaviors.

The intervention is structured over an 8-week period, during which participants are expected to engage daily with the application. The DHT includes several core functionalities:

Digital Sleep Diaries: Participants document their sleep habits daily, including sleep onset latency, total sleep duration, wake after sleep onset, and sleep efficiency. This self-monitoring aims to increase sleep-awareness and encourage consistent engagement with healthy sleep behaviors.

Personalized Educational Content: Users gain access to educational modules designed according to CBT-I principles. Topics include optimizing the sleep environment, maintaining consistent sleep schedules, managing lifestyle factors affecting sleep, and addressing common misconceptions about sleep.

Relaxation and Mindfulness Exercises: The app provides guided audio and video exercises focusing on relaxation techniques such as deep breathing and progressive muscle relaxation, alongside mindfulness practices intended to reduce pre-sleep arousal and facilitate better sleep.

Interactive Chatbot: An integrated conversational agent assists users in navigating app functionalities, provides personalized reminders, motivational feedback, and real-time assistance, enhancing user engagement and compliance.

Participants (N=50) are recruited from the outpatient clinic at Borgo Roma Hospital, Verona. Eligible individuals are randomly assigned in a 1:1 ratio to either receive the DHT intervention combined with Treatment as Usual (DHT + TAU), or Treatment as Usual (TAU) alone. TAU involves standardized educational materials on sleep hygiene practices provided via printed booklets and continued management under the patient's usual healthcare provider.

Assessments are conducted at baseline (T0), immediately post-intervention (T1), and at a 6-month follow-up (T2). Primary outcomes focus on usability and acceptability, measured by the User Experience Questionnaire (UEQ), digital engagement metrics, and adherence to sleep hygiene practices via the Sleep Hygiene Index (SHI). Secondary outcomes assess preliminary efficacy regarding insomnia severity (Insomnia Severity Index - ISI), mood disturbances (Hospital Anxiety and Depression Scale - HADS), and overall health-related quality of life (Short Form Health Survey - SF-12).

Data collection employs the secure LimeSurvey platform to ensure participant confidentiality and data protection according to GDPR standards. Data analysis includes Linear Mixed Effects Models, exploratory analyses for identifying predictors of treatment response, and sensitivity analyses for assessing robustness of findings.

This feasibility trial aims to inform future large-scale studies by evaluating the potential benefits and limitations of using a scalable, non-medical DHT in the routine management of chronic insomnia. Results are anticipated to contribute substantially to the evidence base supporting digital interventions as viable adjuncts to standard care for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years
* Diagnosis of chronic insomnia according to DSM-5 criteria
* Willingness to participate in the study and provide informed consent
* Personal active email address
* Ownership of a compatible mobile device with internet access (for the DHT group)

Exclusion Criteria:

* Medical conditions requiring hospital admission during the study period
* Comorbid diagnosis of sleep-related breathing disorders
* Neurological disorders affecting sleep (e.g., narcolepsy, parasomnias, epilepsy, neurodegenerative diseases)
* Currently receiving psychological treatment for insomnia or planning to do so within the next 6 months
* Incompatible smartphone or lack of internet access (for DHT group)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Usability and Acceptability of Digital Health Technology (DHT) | After 8 weeks of intervention (T1)
  Usability and acceptability measured by the User Experience Questionnaire (UEQ) and digital engagement metrics, including app access frequency, session duration, notification interactions, and drop-out rates.
Adherence to Sleep Hygiene Practices | Baseline (T0), after 8 weeks (T1), and at 6-month follow-up (T2)
  Change in adherence to recommended sleep hygiene behaviors assessed through the Sleep Hygiene Index (SHI).

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline (T0), after 8 weeks (T1), and at 6-month follow-up (T2)
  Change in insomnia severity measured using the Insomnia Severity Index, evaluating subjective sleep disturbance and related daytime impairment.
Mood and Emotional Distress | Baseline (T0), after 8 weeks (T1), and at 6-month follow-up (T2)
  Change in anxiety and depression symptoms assessed using the Hospital Anxiety and Depression Scale (HADS).
Health-Related Quality of Life | Baseline (T0), after 8 weeks (T1), and at 6-month follow-up (T2)
  Change in quality of life across multiple dimensions (e.g., physical functioning, emotional wellbeing) assessed using the Short Form Health Survey (SF-12).

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Borgo Roma - Neurologia B, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will not be shared due to institutional data protection policies and GDPR compliance. Given the sensitivity of health-related personal data and the nature of the digital tools involved, sharing IPD externally poses potential privacy and security risks that cannot be sufficiently mitigated. Additionally, participants were informed that their data would only be accessible to authorized personnel directly involved in the research.

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Watanabe Y, Kuroki T, Ichikawa D, Ozone M, Uchimura N, Ueno T. Effect of smartphone-based cognitive behavioral therapy app on insomnia: a randomized, double-blind study. Sleep. 2023 Mar 9;46(3):zsac270. doi: 10.1093/sleep/zsac270. PMID 36355920
- [Background] Terzano MG, Parrino L, Cirignotta F, Ferini-Strambi L, Gigli G, Rudelli G, Sommacal S; Studio Morfeo Committee. Studio Morfeo: insomnia in primary care, a survey conducted on the Italian population. Sleep Med. 2004 Jan;5(1):67-75. doi: 10.1016/j.sleep.2003.09.006. PMID 14725829
- [Background] Stepanski EJ, Wyatt JK. Use of sleep hygiene in the treatment of insomnia. Sleep Med Rev. 2003 Jun;7(3):215-25. doi: 10.1053/smrv.2001.0246. PMID 12927121
- [Background] Spielman AJ, Caruso LS, Glovinsky PB. A behavioral perspective on insomnia treatment. Psychiatr Clin North Am. 1987 Dec;10(4):541-53. PMID 3332317
- [Background] Shapiro SL, Carlson LE, Astin JA, Freedman B. Mechanisms of mindfulness. J Clin Psychol. 2006 Mar;62(3):373-86. doi: 10.1002/jclp.20237. PMID 16385481
- [Background] Shamim SA, Warriach ZI, Tariq MA, Rana KF, Malik BH. Insomnia: Risk Factor for Neurodegenerative Diseases. Cureus. 2019 Oct 26;11(10):e6004. doi: 10.7759/cureus.6004. PMID 31807391
- [Background] Schuffelen J, Maurer LF, Lorenz N, Rotger A, Pietrowsky R, Gieselmann A. The clinical effects of digital cognitive behavioral therapy for insomnia in a heterogenous study sample: results from a randomized controlled trial. Sleep. 2023 Nov 8;46(11):zsad184. doi: 10.1093/sleep/zsad184. PMID 37428712
- [Background] Riemann D, Espie CA, Altena E, Arnardottir ES, Baglioni C, Bassetti CLA, Bastien C, Berzina N, Bjorvatn B, Dikeos D, Dolenc Groselj L, Ellis JG, Garcia-Borreguero D, Geoffroy PA, Gjerstad M, Goncalves M, Hertenstein E, Hoedlmoser K, Hion T, Holzinger B, Janku K, Jansson-Frojmark M, Jarnefelt H, Jernelov S, Jennum PJ, Khachatryan S, Krone L, Kyle SD, Lancee J, Leger D, Lupusor A, Marques DR, Nissen C, Palagini L, Paunio T, Perogamvros L, Pevernagie D, Schabus M, Shochat T, Szentkiralyi A, Van Someren E, van Straten A, Wichniak A, Verbraecken J, Spiegelhalder K. The European Insomnia Guideline: An update on the diagnosis and treatment of insomnia 2023. J Sleep Res. 2023 Dec;32(6):e14035. doi: 10.1111/jsr.14035. PMID 38016484
- [Background] Riemann D, Spiegelhalder K, Feige B, Voderholzer U, Berger M, Perlis M, Nissen C. The hyperarousal model of insomnia: a review of the concept and its evidence. Sleep Med Rev. 2010 Feb;14(1):19-31. doi: 10.1016/j.smrv.2009.04.002. Epub 2009 May 28. PMID 19481481
- [Background] Riemann D, Nissen C, Palagini L, Otte A, Perlis ML, Spiegelhalder K. The neurobiology, investigation, and treatment of chronic insomnia. Lancet Neurol. 2015 May;14(5):547-58. doi: 10.1016/S1474-4422(15)00021-6. Epub 2015 Apr 12. PMID 25895933
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- [Background] Palagini L, Piarulli A, Menicucci D, Cheli E, Lai E, Bergamasco M, Mauri M, Kyle SD, Espie CA, Gemignani A. Metacognitive beliefs relate specifically to sleep quality in primary insomnia: a pilot study. Sleep Med. 2014 Aug;15(8):918-22. doi: 10.1016/j.sleep.2014.03.017. Epub 2014 May 9. PMID 24916095
- [Background] Ohayon MM. Epidemiology of insomnia: what we know and what we still need to learn. Sleep Med Rev. 2002 Apr;6(2):97-111. doi: 10.1053/smrv.2002.0186. PMID 12531146
- [Background] Ning Y, Teixayavong S, Shang Y, Savulescu J, Nagaraj V, Miao D, Mertens M, Ting DSW, Ong JCL, Liu M, Cao J, Dunn M, Vaughan R, Ong MEH, Sung JJ, Topol EJ, Liu N. Generative artificial intelligence and ethical considerations in health care: a scoping review and ethics checklist. Lancet Digit Health. 2024 Nov;6(11):e848-e856. doi: 10.1016/S2589-7500(24)00143-2. Epub 2024 Sep 17. PMID 39294061
- [Background] Muench A, Vargas I, Grandner MA, Ellis JG, Posner D, Bastien CH, Drummond SP, Perlis ML. We know CBT-I works, now what? Fac Rev. 2022 Feb 1;11:4. doi: 10.12703/r/11-4. eCollection 2022. PMID 35156100
- [Background] Morin CM, LeBlanc M, Daley M, Gregoire JP, Merette C. Epidemiology of insomnia: prevalence, self-help treatments, consultations, and determinants of help-seeking behaviors. Sleep Med. 2006 Mar;7(2):123-30. doi: 10.1016/j.sleep.2005.08.008. Epub 2006 Feb 3. PMID 16459140
- [Background] Mayer G, Jennum P, Riemann D, Dauvilliers Y. Insomnia in central neurologic diseases--occurrence and management. Sleep Med Rev. 2011 Dec;15(6):369-78. doi: 10.1016/j.smrv.2011.01.005. Epub 2011 Apr 9. PMID 21481621
- [Background] Maurer LF, Espie CA, Kyle SD. How does sleep restriction therapy for insomnia work? A systematic review of mechanistic evidence and the introduction of the Triple-R model. Sleep Med Rev. 2018 Dec;42:127-138. doi: 10.1016/j.smrv.2018.07.005. Epub 2018 Sep 1. PMID 30177248
- [Background] Mastin DF, Bryson J, Corwyn R. Assessment of sleep hygiene using the Sleep Hygiene Index. J Behav Med. 2006 Jun;29(3):223-7. doi: 10.1007/s10865-006-9047-6. Epub 2006 Mar 24. PMID 16557353
- [Background] Lorenz N, Heim E, Roetger A, Birrer E, Maercker A. Randomized Controlled Trial to Test the Efficacy of an Unguided Online Intervention with Automated Feedback for the Treatment of Insomnia. Behav Cogn Psychother. 2019 May;47(3):287-302. doi: 10.1017/S1352465818000486. Epub 2018 Sep 6. PMID 30185239
- [Background] Hong JS, Wasden C, Han DH. Introduction of digital therapeutics. Comput Methods Programs Biomed. 2021 Sep;209:106319. doi: 10.1016/j.cmpb.2021.106319. Epub 2021 Jul 29. PMID 34364181
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Espie CA, Kyle SD, Hames P, Gardani M, Fleming L, Cape J. The Sleep Condition Indicator: a clinical screening tool to evaluate insomnia disorder. BMJ Open. 2014 Mar 18;4(3):e004183. doi: 10.1136/bmjopen-2013-004183. PMID 24643168
- [Background] Espie CA, Henry AL. Disseminating cognitive behavioural therapy (CBT) for insomnia at scale: capitalising on the potential of digital CBT to deliver clinical guideline care. J Sleep Res. 2023 Dec;32(6):e14025. doi: 10.1111/jsr.14025. Epub 2023 Aug 29. PMID 37642008
- [Background] Erten Uyumaz B, Feijs L, Hu J. A Review of Digital Cognitive Behavioral Therapy for Insomnia (CBT-I Apps): Are They Designed for Engagement? Int J Environ Res Public Health. 2021 Mar 12;18(6):2929. doi: 10.3390/ijerph18062929. PMID 33809308
- [Background] Darden M, Espie CA, Carl JR, Henry AL, Kanady JC, Krystal AD, Miller CB. Cost-effectiveness of digital cognitive behavioral therapy (Sleepio) for insomnia: a Markov simulation model in the United States. Sleep. 2021 Apr 9;44(4):zsaa223. doi: 10.1093/sleep/zsaa223. PMID 33151330
- [Background] Baek K, Jeong J, Kim HW, Shin DH, Kim J, Lee GH, Cho JW. Seasonal and Weekly Patterns of Korean Adolescents' Web Search Activity on Insomnia: Retrospective Study. JMIR Form Res. 2024 Oct 11;8:e52977. doi: 10.2196/52977. PMID 39311496
- [Background] Castronovo V, Galbiati A, Sforza M, Poletti M, Giarolli L, Kuo T, Zucconi M, Manconi M, Hensley M, Morin C, Ferini-Strambi L. Long-term clinical effect of group cognitive behavioral therapy for insomnia: a case series study. Sleep Med. 2018 Jul;47:54-59. doi: 10.1016/j.sleep.2018.03.017. Epub 2018 Apr 11. PMID 29753926
- [Background] Baglioni C, Altena E, Bjorvatn B, Blom K, Bothelius K, Devoto A, Espie CA, Frase L, Gavriloff D, Tuuliki H, Hoflehner A, Hogl B, Holzinger B, Jarnefelt H, Jernelov S, Johann AF, Lombardo C, Nissen C, Palagini L, Peeters G, Perlis ML, Posner D, Schlarb A, Spiegelhalder K, Wichniak A, Riemann D. The European Academy for Cognitive Behavioural Therapy for Insomnia: An initiative of the European Insomnia Network to promote implementation and dissemination of treatment. J Sleep Res. 2020 Apr;29(2):e12967. doi: 10.1111/jsr.12967. Epub 2019 Dec 19. PMID 31856367
- [Background] American Psychiatric Association (2013). Manuale diagnostico e statistico dei disturbi mentali - Quinta edizione. DSM-5. Tr.it. Raffaello Cortina, Milano, 2015.